CLINICAL TRIAL: NCT01169350
Title: A Phase 2 Study of Positron Emission Tomography Imaging With [18F]-Fluoromisonidazole (FMISO) and [18F]-Fluorodeoxyglucose (FDG) for Assessment of Tumor Hypoxia in Soft Tissue Sarcoma
Brief Title: 18F-Fluoromisonidazole and Fludeoxyglucose F 18 PET/CT Patients With Soft Tissue Sarcoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: funding source ended earlier than anticipated
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NCI-2011-01442; NCI-2011-01442 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 8468; CDR0000665359; UW-8468; 6971 (Other: University of Washington Medical Center); 8468 (Other: CTEP); N01CM37008-9-0-0 (NIH)
Record Dates: First submitted 2010-07-23; First posted 2010-07-26 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Recurrent Adult Soft Tissue Sarcoma; Stage I Adult Soft Tissue Sarcoma; Stage II Adult Soft Tissue Sarcoma; Stage III Adult Soft Tissue Sarcoma; Stage IV Adult Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Fluorodeoxyglucose F18; fluoromisonidazole; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (18F FDG and 18F FMISO PET/CT) (Experimental): Patients undergo 18F FDG and 18F FMISO PET/CT scans before starting neoadjuvant chemotherapy (without or without radiotherapy) and after completion of 4 courses of neoadjuvant therapy.
  Interventions: Radiation: fludeoxyglucose F 18; Other: 18F-fluoromisonidazole; Procedure: positron emission tomography; Procedure: computed tomography; Other: laboratory biomarker analysis

INTERVENTIONS:
Radiation: fludeoxyglucose F 18 — Undergo 18F FDG and 18F FMISO PET/CT scans
Other: 18F-fluoromisonidazole — Undergo 18F FDG and 18F FMISO PET/CT scans
Procedure: positron emission tomography — Undergo 18F FDG and 18F FMISO PET/CT scans
Procedure: computed tomography — Undergo 18F FDG and 18F FMISO PET/CT scans
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying 18F-fluoromisonidazole and fludeoxyglucose F 18 PET/CT scans to see how well they work in assessing oxygen in tumor tissue of patients with soft tissue sarcoma undergoing chemotherapy with or without radiation therapy. Using diagnostic procedures, such as 18F-fluoromisonidazole and fludeoxyglucose F 18 PET scan and CT scan, to find oxygen in tumor cells may help in planning cancer treatment. It may also help doctors predict how well a patient will respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the potential of 18F-fluoromisonidazole ([18F] FMISO) as a non-invasive indicator of tissue hypoxia to provide tumor-imaging data that correlates with tissue markers of hypoxia in patients with soft tissue sarcoma treated with neoadjuvant chemotherapy with or without radiotherapy.

SECONDARY OBJECTIVES:

I. Test [18F] FMISO tumor uptake as an independent predictor of patient outcome and if it provides additional predictive power over fludeoxyglucose F 18 PET scan.

II. Test [18F] FMISO tumor uptake as a predictor of response in the subgroup of patients treated with radiotherapy and chemotherapy.

III. Test the reproducibility of [18F] FMISO uptake in tumors by imaging the same patients on sequential days in a test-retest protocol.

IV. Determine the relationship between hypoxia-related biomarkers (HIF1-a and VEGF), proliferation biomarkers (microvascular density, p53, and Ki-67), and regional [18F] FMISO uptake in tumor.

OUTLINE:

Patients undergo fludeoxyglucose F 18 [18F] FDG and 18F-fluoromisonidazole ([18F] FMISO) positron emission tomography (PET)/CT scans before starting neoadjuvant chemotherapy (without or without radiotherapy) and after completion of 4 courses of neoadjuvant therapy.

NOTE: Some patients may undergo repeat [18F] FMISO PET/CT scan within 48 hours after the first [18F] FMISO scan to evaluate the variability (test-retest) of this imaging measurement.

Blood samples are collected after completion of [18F] FMISO and [18F] FDG PET/CT scans for laboratory biomarker studies by IHC assays. Tumor samples from biopsy or surgery are also collected for biomarker studies.

After completion of study procedures, patients are followed up periodically for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed intermediate- or high-grade soft tissue sarcoma

  * Biopsy proven or highly suspicious primary or recurrent disease
  * Tumor size ≥ 2 cm
* Scheduled to undergo neoadjuvant chemotherapy with or without radiotherapy
* Life expectancy ≥ 12 months
* Negative pregnancy test
* Willing to undergo PET scanning
* Willing to undergo possible urinary bladder catheterization (for patients with pelvic or proximal thigh tumors)
* Able to lie on the imaging table for up to 1.5 hours
* Weight ≤ 400 lbs
* Not pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-02; Primary Completion 2011-10 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Eary, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diagnostic (18F FDG and 18F FMISO PET/CT)
Started | 8
Completed | 3
Not Completed | 5
Not completed — Physician Decision | 3
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Received Baseline FDG PET and FMISO PET
Arm/Group | Diagnostic (18F FDG and 18F FMISO PET/CT)
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 61 [45 to 80]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline Hypoxic Volume (HV)
Description: ANOVA and Kruskal-Wallis analysis will be performed across the different categories to look for significant associations.
Time Frame: Baseline and up to 2 years
Population: Study ended with 8 patients imaged at baseline and only 3 patients had 18F FMISO following therapy.
Measure: Mean (Standard Deviation); unit: Cm^3
Arm/Group | Diagnostic (18F FDG and 18F FMISO PET/CT)
Number analyzed (Participants) | 3
Cm^3 | 9.7 (11.7)

2. Secondary Outcome: Overall Survival
Description: Multivariate Cox regression will be used. The outcome is binary and generalized linear models and logistic regression will be employed.
Time Frame: Up to 2 years
Population: Study ended. No patients were assessed for overall survival.No data were collected for this assessment.
Arm/Group | Diagnostic (18F FDG and 18F FMISO PET/CT)
Number analyzed (Participants) | 0

3. Secondary Outcome: Disease Free Survival
Description: Multivariate Cox regression will be used.
Time Frame: From start of treatment to the follow-up review where recurrent disease is first detected, assessed up to 2 years
Population: Study ended. No patients were assessed for disease free survival.No data were collected for this assessment
Arm/Group | Diagnostic (18F FDG and 18F FMISO PET/CT)
Number analyzed (Participants) | 0

4. Secondary Outcome: Response to Radiation Therapy (XRT) by RECIST Criteria
Description: Will be approached using multivariate logistic regression.
Time Frame: Up to 2 years
Population: Study ended. No patients were assessed for response to radiation therapy (XRT) by RECIST criteria. No data were collected for this assessment.
Arm/Group | Diagnostic (18F FDG and 18F FMISO PET/CT)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected 24hr +/- 4 hours after each administration of [18F] FMISO.
Arm/Group | Diagnostic (18F FDG and 18F FMISO PET/CT)
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less